CLINICAL TRIAL: NCT02689518
Title: Clinical and Genetic Assessment of Treatment Response in Patients With Age-related Macular Degeneration Using Intravitreal Aflibercept Injection
Brief Title: EAGLE: Evaluating Genotypes Using Intravitreal Aflibercept Injection
Acronym: EAGLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Michael Goldbaum, MD, Professor of Ophthalmology in Residence, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EAGLE
Record Dates: First submitted 2014-04-21; First posted 2016-02-24 (Estimated); Results first posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Macular Degeneration; Wet Macular Degeneration
Keywords: AMD; Wet AMD; Macular degeneration; Wet macular degeneration; Neovascularization; Retina; Retinal degeneration
MeSH Terms: conditions — Macular Degeneration; Wet Macular Degeneration; Neovascularization, Pathologic; Retinal Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment - On-Label (Other): On-label intravitreal aflibercept (Eylea) injection 2 mg (0.05 mL) administered every 4 weeks for the first 3 months, followed by 2 mg (0.05 mL) intravitreal injection once every 8 weeks (2 months) with the option to treat monthly based on retreatment criteria for a total duration of 12 months
  Interventions: Drug: Intravitreal aflibercept injection

INTERVENTIONS:
Drug: Intravitreal aflibercept injection — Intravitreal aflibercept injection 2 mg (0.05 mL) administered every 4 weeks for the first 3 months, followed by 2 mg (0.05 mL) intravitreal injection once every 8 weeks(2 months) with the option to treat monthly based on retreatment criteria for a total duration of 12 months.
  Other Names: Eylea

SUMMARY:
Clinical and genetic evaluation of individuals treated with intravitreal aflibercept injection (Eylea) for neovascular age-related macular degeneration (wet AMD)

DETAILED DESCRIPTION:
Clinical and genetic assessment of treatment response in patients with age-related macular degeneration using intravitreal aflibercept injection. This study seeks to determine if different genetic polymorphisms of vascular endothelial growth factor A (VEGF-A) and HtrA serine peptidase 1(HTRA1) and other genes correlate to the response to intravitreal aflibercept injection therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 years
2. Naïve neovascular wet-AMD (has not received treatment before)
3. Willing and able to comply with clinic visits and study-related procedures
4. Provide signed informed consent

Exclusion Criteria:

1. Previous therapy in study eye for AMD or other retinal disease which may be used in the treatment of AMD
2. Previous subfoveal focal laser photocoagulation involving the foveal center in the study eye
3. History of vitrectomy, submacular surgery, or other surgical intervention for AMD in the study eye
4. Any concurrent intraocular condition in the study eye (e.g. diabetic retinopathy or glaucoma) that, in the opinion of the investigator, could either 4.1 require medical or surgical intervention during the study period to prevent or treat visual loss that might result from that condition, or 4.2 if allowed to progress untreated, could likely contribute to loss of at least 2 Snellen equivalent lines of best corrected visual acuity over the study period
5. Active intraocular inflammation (grade trace or above) in the study eye, or history of idiopathic or autoimmune-associated uveitis in either eye
6. Current vitreous hemorrhage in the study eye
7. History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye
8. Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
9. Aphakia, ACIOL, or unstable PCIOL
10. Uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥30 mmHg despite treatment with anti-glaucoma medication)
11. Pregnant or breast-feeding women
12. Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly)
13. Any other condition that the investigator believes would pose a significant hazard to the patient if the investigational therapy were initiated *Contraception is not required for men with documented vasectomy. **Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child bearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Goldbaum, M.D., Principal Investigator — UCSD
Locations (1):
- Shiley Eye Center, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The record for one participant was lost so we will report on 49/50.
Period: Overall Study
Arm/Group | Treatment - On-Label
Started | 49
Completed | 46
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: The record for one participant was lost we will report on 49/50
Arm/Group | Treatment - On-Label
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Anatomic Response
Description: The primary endpoint in the study is the correlation of CFH, HTRA1, VEGFA, C3, TIMP3, APOE, CETP, LIPC, TGFBR1, CFI, and CFB allele frequencies and VEGA expression in lymphoblastoid cell lines with response to intravitreal aflibercept injection treatment, based on anatomic outcomes:
  Early response (at Month 3) - o On optical coherence tomography(SD-OCT)
  * Reduction in central retinal thickness by ≥ 50%, OR
  * Central retinal thickness <300 um, OR
  * Absence of retinal fluid
  Later response (at Month 12) -
  o On SD-OCT
  * Reduction in central retinal thickness by ≥ 50%, OR
  * Central retinal thickness < 300 um, OR
  * Absence of retinal fluid
  Poor response, defined as no reduction of fluid or central retinal thickness at Month 12.
Time Frame: 12 Months
Population: Principal Investigator is no longer associated with the institution. All efforts were exhausted to obtain the data but no data could be found.
Arm/Group | Treatment - On-Label
Number analyzed (Participants) | 0

2. Secondary Outcome: Visual/Treatment Response
Description: The secondary endpoints are a correlation of CFH, VEGF, HTRA1, VEGFA, C3, TIMP3, APOE, CETP, LIPC, TGFBR1, CFI, and CFB allele frequencies:
  With visual outcomes -
  * Early response, defined as a gain ≥ 0 letters at Month 3
  * Later response, defined as a gain ≥ 0 letters at Month 12
  * Poor response, defined as loss of visual acuity (gain <0 letters) at Month 12
  With change in characteristics on fluorescein angiography and fundus photography (lesion size, lesion type, etc)
  With number of injections through Month 12
  o Mean number of intravitreal aflibercept injections required through Month 12 will be calculated for the group overall, and separately by response group (early, later, and no response to treatment).
Time Frame: 12 Months
Population: as for outcome 1
Arm/Group | Treatment - On-Label
Number analyzed (Participants) | 0

3. Other Pre Specified Outcome: Safety - Incidence and Severity of Ocular and Non-ocular Adverse Events
Description: Incidence and severity of ocular and non-ocular adverse events using Aflibercept intravitreal injections will also be evaluated.
Time Frame: 12 Months
Population: as for outcome 1
Arm/Group | Treatment - On-Label
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Principal Investigator is no longer associated with the institution. All efforts were exhausted to obtain the data but no data could be found.
Arm/Group | Treatment - On-Label
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Principal Investigator is no longer associated with the institution. All efforts were exhausted to obtain the data but no data could be found.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-02-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT02689518/Prot_000.pdf